CLINICAL TRIAL: NCT07203482
Title: A Single-center Observational Study of Clinical Outcomes of Clinically Localized Prostate Cancer Undergoing HIFU Therapy
Brief Title: Clinical Outcomes in Prostate Cancer Patients Undergoing HIFU Ablation
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 23-01458
Record Dates: First submitted 2025-09-23; First posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prostate Cancer Patients Scheduled for HIFU Procedure: Participants will be actively followed up for the first 3 years. After that once a year for life, unless they withdraw from the study or no longer seek standard of care at NYU Langone Health.

SUMMARY:
Many reports of clinical outcomes following treatment of localized prostate cancer suffer from lack of prospective long-term data using objective and validated outcome instruments. The purpose of this research database is to prospectively collect data to assess treatment related complications, oncologic outcomes and urinary/sexual function, and identify predictors of complications, oncological control and functional outcomes after Hhigh-intensity focused ultrasound (HIFU) ablation of prostate cancer with the intent to guide further research and improve patient care. We will include subjects who will have a HIFU procedure performed from all Sub-Investigators included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Males, ages 40-95
* Evidence of focal prostate cancer confined to the prostate based on MRI imaging and prostate biopsy
* Patients with clinically localized prostate cancer (no evidence for or concern for metastatic spread of cancer outside of the prostate) that select focal HIFU prostate ablation as their treatment option will be offered inclusion into this prospective data collection research database.
* Patients who have early (Gleason 6 or 7), low grade cancer that is confined to the prostate.
* Willing and able to provide consent.

Exclusion Criteria:

* Patients that are not diagnosed with prostate cancer.
* Patients that are diagnosed with clinically localized prostate cancer, but select other tratment options as their desired treatment.
* Patients that are not willing or are not able to give consent.

Ages: 40 Years to 95 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males, age 40-95 who are prostate cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2050-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Prostate-Specific Antigen (PSA) Levels | Baseline (pre-HIFU ablation procedure), Month 3, Month 6, Month 12, Month 18, Month 24, Month 30, Month 48, Month 60
Change in Urinary Function Score | Baseline (pre-HIFU ablation procedure), Month 3, Month 6, Month 12, Month 18, Month 24, Month 30, Month 48, Month 60
  Urinary Function is assessed using an 8-item questionnaire; each item is rated on a question-specific Likert scale. The total score is the sum of responses and ranges from 0 - 41; lower scores indicate greater urinary function.
Change in Urinary Continence Score | Baseline (pre-HIFU ablation procedure), Month 3, Month 6, Month 12, Month 18, Month 24, Month 30, Month 48, Month 60
  Urinary Continence is assessed using an 2-item questionnaire; each item is rated on a Likert scale from 0-3. The total score is the sum of responses and ranges from 0 - 6; higher scores indicate greater urinary continence.
Change in Sexual Function Score | Baseline (pre-HIFU ablation procedure), Month 3, Month 6, Month 12, Month 18, Month 24, Month 30, Month 48, Month 60
  Sexual Function is assessed using a 6-item questionnaire; each item is rated on a question-specific Likert scale. The total score is the sum of responses and ranges from 0 - 29; lower scores indicate greater sexual function.
Change in Ejaculatory Function Score | Baseline (pre-HIFU ablation procedure), Month 3, Month 6, Month 12, Month 18, Month 24, Month 30, Month 48, Month 60
  Ejaculatory Function is assessed using a 4-item questionnaire; each item is rated on a question-specific Likert scale. The total score is the sum of responses and ranges from 1 - 20; higher scores indicate greater ejaculatory function.
Change in Sexual Health Inventory for Men (SHIM) Score | Baseline (pre-HIFU ablation procedure), Month 3, Month 6, Month 12, Month 18, Month 24, Month 30, Month 48, Month 60
  SHIM is a 5-item questionnaire assessing sexual health in men; each item is rated on a question-specific Likert scale. The total score is the sum of responses and ranges from 1-20; higher scores indicate greater sexual health.
Decision Regret Score | Month 3, Month 6, Month 12, Month 18, Month 24, Month 30, Month 48, Month 60
  Regret toward receiving HIFU ablation focal therapy is assessed using a 5-item questionnaire. Each item is rated on a Likert scale from 1-5; the total score is the sum of responses and ranges from 5-25. Lower scores indicate less regret with the decision.
Number of Participants with Persistence or Recurrence of Cancer within the Treatment Zone on Post-Treatment Imaging | Up to Month 60
Number of Participants with New Lesions in the Non-Treated Prostate on Post-Treatment Imaging | Up to Month 60
Number of Participants with Persistence or Recurrence of Cancer within the Treatment Zone on Post-Treatment Prostate Biopsy | Up to Month 60
Number of Participants with New Lesions in the Non-Treated Prostate on Post-Treatment Prostate Biopsy | Up to Month 60

CONTACTS AND LOCATIONS:
Overall Officials: James Wysock, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - NYU Langone Health - Cobble Hill, Brooklyn, New York
  - NYU Langone Health - Tisch Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset will be shared upon reasonable request beginning 9 to 36 months after publication or as required by a condition of awards or supporting agreements, provided the requesting investigator executes a data use agreement with NYU Langone Health. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's Data Sharing Strategy Board (DSSB). Requests should be directed to: James.Wysock@nyulangone.org. The protocol and statistical analysis plan will be posted on Clinicaltrials.gov only as required by federal regulation or supporting awards and agreements.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to James.Wysock@nyulangone.org. To gain access, data requestors will need to sign a data access agreement. This instance of data sharing will also require separate IRB review as well as review from NYU Langone's DSSB.